CLINICAL TRIAL: NCT02818075
Title: Mobile Phone Based Peer Support to Prevent Postpartum Depression Among Adolescent Mothers: A Pilot Randomized Controlled Trial
Brief Title: Mobile Phone Based Peer Support to Prevent Postpartum Depression Among Adolescent Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Barbara Chyzzy, PhD Candidate, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 32189
Record Dates: First submitted 2016-06-06; First posted 2016-06-29 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Postpartum Depression
Keywords: Peer support; Postpartum Depression; Adolescent Pregnancy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Phone Based Peer Support (Experimental): Mobile phone-based peer support (MPPS)
  Interventions: Other: Mobile Phone Based Peer Support; Other: Usual Care
- Usual Care (Active Comparator): Standard community prenatal and postpartum support services
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Mobile Phone Based Peer Support — Adolescents allocated to the experimental group will have access to all standard prenatal and postpartum community supports. In addition, mobile phone-based peer support (MPPS), which consists of support provided by a peer mentor via mobile phone (with both voice calling and Short Message Service text message capabilities) will be provided during pregnancy and for 12 weeks postpartum. Peer support is defined as a specific type of social support (informational, appraisal, and emotional support) that is provided by a peer mentor who possesses experiential knowledge of adolescent motherhood and is of similar age to the participant.
  Arms: Mobile Phone Based Peer Support
Other: Usual Care — Participants allocated to the usual care group will not receive the peer support intervention but will have access to all standard community prenatal and postpartum support services such as 1) the Canada Prenatal Nutrition Program; 2) postpartum home visits / telephone support from a public health nurse; 3) postpartum appointments with midwives, obstetrician, family physician, and / or pediatricians, and 4) prenatal and postpartum support as needed from psychiatrists, psychologists, social workers, breastfeeding clinics, and community resources.

SUMMARY:
This pilot study will evaluate the feasibility and acceptability of a mobile phone based peer support intervention among adolescent mothers. Half of the participants will receive usual care plus the peer support intervention and the other half of the participants will receive usual care only.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is one of several postpartum mood disorders and is classified as a major depressive disorder. It has the highest inception rate during the first 12 weeks postpartum and is frequently comorbid with anxiety disorders or significant anxiety symptoms. PPD is the most frequent form of maternal morbidity following childbirth and has serious negative consequences including maternal suffering, impaired maternal-infant interactions and cognitive, behavioural and emotional problems in infants and children. As a result of these negative consequences, PPD has been deemed a major public health concern warranting preventive intervention. Adolescent mothers are a particularly vulnerable maternal population who are at approximately three times greater risk for developing postpartum depression (PPD) compared to adult mothers, with an estimated prevalence of 38%. In 2011, over 65,000 live births were recorded to adolescents between 15-24 years of age in Canada, which represents a significant number of mothers at risk for developing PPD.

Several variables have been identified as predictors for PPD among adolescent mothers; however, the one variable which has been consistently identified in studies is a lack of social support. A detailed analysis of social support variables in predictive studies among adolescent mothers clearly identifies not having someone to talk with about their problems as a major deficiency in social support. These findings are not surprising as the relationship between lack of social support and reduced psychological well-being has been well established. Evidence shows that decreased social network size, fewer close relationships, and lower perceived adequacy of social support are all linked to depressive symptomatology.

Peer to peer support, a form of social support, has been shown to improve health outcomes in various age groups including adolescents. Peers are lay individuals who have similar characteristics and experiences as a target population and can share pragmatic knowledge and empathic understanding. The provision of peer support includes (a) informational support (knowledge, facts, and suggestions), (b) emotional support (attentive listening, caring and reassurance) and (c) appraisal support (motivation, encouragement and positive communication) which is delivered by a peer.

The purpose of this study is to evaluate the feasibility and acceptability of a mobile phone-based peer support intervention and adherence with the trial protocol to inform a future definitive full-scale randomized controlled trial.

The design is a pilot randomized controlled trial. Forty eligible and consenting pregnant adolescents age 16-24 years will be randomized into an intervention or control group. Adolescents in the control group will receive standard prenatal and postpartum in-hospital and community care. Adolescents in the intervention group will receive the same standard care as the control group plus a mobile phone-based peer support intervention. Mobile phone-based peer support will consist of support provided by a trained peer mentor starting in the participant's last trimester of pregnancy and continuing for 12 weeks postpartum. Peer mentors are young mothers between 16-24 years of age who will receive 12 hours of training to learn how to provide support to new young mothers. Peer support will be provided either via voice calling or text messaging depending on the participant's preference. Additionally, acceptability by participants the intervention group will be evaluated via questionnaire and semi-structured interview to determine likes/dislikes and areas for improvement. Preliminary effectiveness will be a secondary outcome with depressive and anxiety symptoms measured using the Edinburgh Postnatal Depression Scale and the Speilberger State Anxiety Inventory at 12 weeks postpartum. Social support and health services utilization will also be measured at 12 weeks postpartum.

This study will provide evidence about a novel approach to preventing PPD among adolescent mothers. Results will reveal which components of peer support (informational, emotional or appraisal support) and which aspects of mobile phone technology (voice-calling, text messaging or a combination of both) are most acceptable for adolescent mothers. Based on the results of this current study, new knowledge will be gained in relation to the provision of peer support among adolescent mothers using mobile technology. This trial will provide valuable information to address a major public health concern (PPD) in a highly vulnerable population (adolescent mothers).

ELIGIBILITY:
Inclusion Criteria:

* > 16 years and < 24 years
* > 28 weeks gestation (third trimester of pregnancy)
* Singleton pregnancy
* Able to speak, read and understand English

Exclusion Criteria:

* Edinburgh Postnatal Depression Scale (EPDS) score > 12
* High risk pregnancy (such as placenta previa, placental abruption, unmanaged pre-eclampsia, intrauterine growth restriction, or known fetal abnormality)
* Current substance use during pregnancy (such as alcohol, cocaine, hallucinogens, marijuana, methadone treatment, narcotics, opioids, etc)
* Active psychosis, schizophrenia, or bipolar disorder
* Adolescents who are subject to a Child Protection Order or who are in foster care.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01-21 (Actual); Study Completion 2018-01-21 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the Participant Eligibility Assessment Form | Through to study completion (12 weeks postpartum)
  The Participant Eligibility Assessment Form will be completed by the PI and used to determine 1) recruitment procedures (effectiveness of recruitment approaches, recruitment rate and reasons for non-participation), 2) screening procedures (appropriateness of inclusion and exclusion criteria), and 3) randomization (willingness to be randomized).
Acceptability as assessed by the validated Peer Support Evaluation Inventory | 12 weeks postpartum
  Acceptability will assessed using the validated Peer Support Evaluation Inventory and will describe maternal perspectives of the Mobile Phone Based Peer Support intervention and will be measured at 12 weeks postpartum
Compliance as assessed by the Activity Log Form | Through to study completion (12 weeks postpartum)
  Adherence-related measures include 1) the number of first contacts (three-way contact) initiated by the PI between the participant and the peer mentor within 72 hours post randomization; 2) the number of Activity Logs completed electronically by the peer mentor compared to the number of contacts made between the peer mentor and the participant; 3) the degree of intervention fidelity measured by the number of Activity Logs completed in congruence between the PI and peer mentors and 4) the number of participants who complete outcomes measures at 12 weeks postpartum.
Support strategies as assessed by the Activity Log Form | Through to study completion (12 weeks postpartum)
  The Activity Log will be used to determine 1) type of support strategies implemented (informational, emotional or appraisal support); 2) type of contact (text-message, voice-call or face to face meeting); 3) dosage (number of voice calls and text messages; duration of contact with peer mentor); 4) technical issues related to the mobile phones and data plans; 5) issues related to participant safety; and 6) whether calls/texts were initiated by the participant or peer mentor intervention is able to be implemented

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 12 weeks postpartum
  To measure depressive symptomatology
State-Trait Anxiety Inventory (STAI) | 12 weeks postpartum
  To measure anxiety levels
Short Form Social Support Questionnaire (SSQ6) | 12 weeks postpartum
  To measure levels of social support since delivery of participant's baby
Health Services Utilization Questionnaire | 12 weeks postpartum
  To collect data on complications during delivery, health service utilization since delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No